CLINICAL TRIAL: NCT02122692
Title: Interventional, Open-label, One-sequence Crossover Study to Evaluate the Effect of Multiple Doses of Itraconazole (Inhibitor of CYP3A4/5) on the Multiple Dose Pharmacokinetics of Lu AE58054 in Healthy Subjects
Brief Title: Effect of Multiple Doses of Itraconazole on the Multiple Dose Pharmacokinetics of Lu AE58054 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15820A; 2013-003597-27 (EudraCT Number)
Record Dates: First submitted 2014-04-23; First posted 2014-04-24 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — (2-(6-fluoro-1H-indol-3-yl)-ethyl)-(3-(2,2,3,3-tetrafluoropropoxy)benzyl)amine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lu AE58054 30 mg + itraconazole 200 mg (Experimental)
  Interventions: Drug: Lu AE58054 30 mg; Drug: Lu AE58054 30 mg + itraconazole 200 mg; Drug: Itraconazole

INTERVENTIONS:
Drug: Lu AE58054 30 mg — Lu AE58054 encapsulated film-coated tablets, once daily, Day 1-5, orally
Drug: Lu AE58054 30 mg + itraconazole 200 mg — Lu AE58054 encapsulated film-coated tablets, once daily, Day 6-11, orally + itraconazole capsules, once daily, Day 6-11, orally
Drug: Itraconazole — Itraconazole capsules, once daily, Day 12-13, orally

SUMMARY:
To examine the effect of the strong CYP3A4/5 inhibitor itraconazole (200 mg QD) on the multipledose exposure of Lu AE58054 (30 mg QD) in healthy subjects (CYP2D6 extensive metabolisers).

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion into the study if they meet each of the following criteria:

* Men and women, aged 18 - 45 years.
* Body weight at least 50 kg and Body Mass index 19 - 28 kg/m2.
* Good general health ascertained by a detailed medical history, laboratory tests and physical examination.
* Non-childbearing potential or use of contraception (both sexes).
* Women must not be pregnant or lactating.
* Known CYP2D6 genotype (Extensive metaboliser (n=15) and poor metaboliser (n =5)) .

Other Inclusion and Exclusion Criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the Lu AE58054 plasma concentration-time curve from time zero to 24 hours post-dose (AUC0-24) | Day 5 and Day 11
Maximum observed concentration (Cmax) of Lu AE58054 | Day 5 and Day 11

SECONDARY OUTCOMES:
Plasma pharmacokinetics for Lu AE58054: AUC0-24, Cmax, time at which maximum observed plasma concentration occurred (tmax), apparent oral clearance (CL/F), half life (t½) and apparent volume of distribution Vz/F | Day 5 and Day 11
Plasma pharmacokinetics for relevant metabolites: AUC0-24, Cmax, tmax, t½ and metabolic ratio (MR) | Day 5 and Day 11
Plasma pharmacokinetic parameters for itraconazole: CTrough | Day 6 to Day 13
Adverse events | Up to Day 18, including a safety follow-up
Columbia Suicide Severity Rating Scale (C-SSRS) categorization based on Columbia Classification Algorithm of Suicide Assessment (C-CASA) definitions | Up to Day 18, including a safety follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- FR801, Rennes, France